CLINICAL TRIAL: NCT05974787
Title: Identification of Potential Improvements in the Acute Care Pathway for Cancer Patients in the Emergency Department (OVERSEE - I Trial)
Brief Title: Potential Improvements in the Pre-emergency Department Care for Cancer Patients
Acronym: OVERSEE-I
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Jason den Duijn, Principal Investigator, Erasmus Medical Center
Other Study IDs: 10841
Record Dates: First submitted 2023-07-18; First posted 2023-08-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-08

CONDITIONS: Cancer; Emergencies
MeSH Terms: conditions — Neoplasms; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cancer patients: All adult patients with solid or hematological malignancies and receiving systemic therapy or having received systemic therapy within the last 3 months admitted to the emergency department of the Erasmus Medical Center for the oncology, hematology, lung- and neuro-oncology medical unit are eligible for inclusion.
  Interventions: Behavioral: Emergency department cancer patients interview

INTERVENTIONS:
Behavioral: Emergency department cancer patients interview — The interview focuses on several parts of the (pre-)admission process: The first part is regarding the barriers and facilitators encountered during the (pre-)admission process. The second part will focus on the timeline that led to an emergency department (ED) visit. It will be established when and which symptoms were first detected. The third part is regarding the number and type of health care workers that were contacted before visiting the ED. The fourth part will be about the actions and considerations taken before the ED visit.

SUMMARY:
The goal of this single center prospective cross-sectional study is to identify the facilitators and barriers in the course of the disease that starts when symptoms first arise until patients with solid and hematologic malignancies arrive in the emergency department (ED). The main question it aims to answer are: Is there a potential relation between the lag-time and the ED length of stay (LOS) and the chance of admission. Participants will be asked to participate in a one-time interview, that focusses on the pre-admission process.

DETAILED DESCRIPTION:
The goal of this single center prospective cross-sectional study is to identify the facilitators and barriers in the course of the disease that starts when symptoms first arise until patients with solid and hematologic malignancies arrive in the emergency department (ED). The main question it aims to answer are: Is there a potential relation between the lag-time and the emergency department length of stay and the chance of admission. Participants will be asked to participate in a one-time interview, that focusses on the pre-admission process. The interview focuses on several parts of the (pre-)admission process: The first part is regarding the timeline that led to an ED visit. The investigators will establish, when and which symptoms were first detected. The second part are regarding the number and type of health care workers that were contacted before visiting the ED. The third part will be about the actions that were taken before the ED visit.

ELIGIBILITY:
Inclusion criteria:

* Patients with solid or hematological malignancies and receiving systemic therapy or having received systemic therapy within the last 3 months.
* Presented at or admitted from the emergency department for the oncology, hematology, neuro- or lung-oncology clinical unit.
* Awake and conscious.
* Possible to answer questions within 48 hours after presentation at the emergency department (ED).

Exclusion Criteria:

* <18 years old
* Only received a surgical intervention as cancer treatment
* Admitted to the ED for the surgical department
* Not willing or able to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the emergency department (ED) of Erasmus medical center (MC) yearly around 1600 patients with cancer are presented to the ED. Based on the study design we will conduct interviews with 75 to 100 patients with solid and hematologic malignancies, who are receiving systemic therapy or have received systemic therapy within the last 3 months and are admitted to the ED department of the Erasmus MC for the oncology, hematology, lung- and neuro-oncology medical unit. If present, the interview will also be held with the family caregiver.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Clusters of facilitators experienced by cancer patients. | Through study completion, an average of 6 months
  Different (sub)clusters of facilitators experienced by cancer patients visiting the emergency department (ED)
clusters of barriers experienced by cancer patients. | Through study completion, an average of 6 months
  Different (sub)clusters of barriers experienced by cancer patients visiting the ED

SECONDARY OUTCOMES:
Time-to-speak | Through study completion, an average of 6 months
  The time between the first notice of symptoms and the first time these complaints were spoken out to the primary giver
Time-to-contact | Through study completion, an average of 6 months
  The time between the first time complaints are spoken out and contact is made with a healthcare professional
Time-to-present | Through study completion, an average of 6 months
  The time between the first contact with a healthcare professional and the presentation at the ED
Difference in group average lag-time between day, evening and night | Through study completion, an average of 6 months
  Difference in group average lag-time between day, evening and night
Difference in group average lag-time between weekdays (Monday 08:00 till Friday 23:59) and weekend (Saturday 00:00 and Monday 7:59) | Through study completion, an average of 6 months
  Difference in group average lag-time between weekdays (Monday 08:00 till Friday 23:59) and weekend (Saturday 00:00 and Monday 7:59)
Correlation between number of contacted healthcare providers before presentation at the ED and the lag- time. | Through study completion, an average of 6 months
  Correlation between number of contacted healthcare providers before presentation at the ED and the lag- time.
Willingness to participate | Through study completion, an average of 6 months
  the percentage of people that participated in this study in comparison to the people approached for this study.
Lag-time | Through study completion, an average of 6 months
  The time between the first onset of symptoms and a visit to the ED.
ED length of stay (LOS) | Through study completion, an average of 6 months
  The time a patient spends in the ED
Disposition | Through study completion, an average of 6 months
  The outcome of a visit to the ED, being either admission or home
Patient characteristics | Through study completion, an average of 6 months
  Age, sex, type of cancer, type of complaint, triage category, number of prior visits
Correlation between lag-time and ED-LOS | Through study completion, an average of 6 months
  Correlation between lag-time and ED-LOS
Correlation between lag-time and disposition | Through study completion, an average of 6 months
  Correlation between lag-time and disposition
Correlation between lag-time and patient characteristics | Through study completion, an average of 6 months
  Correlation between lag-time and patient characteristics
ED crowding | Through study completion, an average of 6 months
  Measure of business of the ED, composed of the number of patients in the ED and the color coding used for crowding

CONTACTS AND LOCATIONS:
Overall Officials: Jason den Duijn, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No